CLINICAL TRIAL: NCT05351047
Title: A Phase I, Randomized, Single-blind, Placebo-controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD2373 Following Multiple Ascending Dose Administration to Healthy Male Participants of Sub-Saharan West African Ancestry
Brief Title: A Study to Assess Safety, Tolerability, PK and PD of AZD2373 in Healthy Male Participants of Sub-Saharan West African Ancestry
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: D6800C00002
Record Dates: First submitted 2022-04-01; First posted 2022-04-28 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Healthy Volunteers
Keywords: Phase 1; Randomized; Single-blind; Placebo controlled; AZD2373; Multiple Ascending Dose

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This study is single-blind (in which the study center staff remain blinded during the clinical conduct of a given cohort) with regard to treatment (AZD2373 or placebo) at each dose level. Study participants will be blinded to treatment allocation throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): Once weekly dosing for 4 weeks (Dosing Days 1, 8, 15 and 22) OR Once weekly dosing for 6 weeks (Dosing Days 1, 8, 15, 22, 29 and 36) randomized subjects will receive a subcutaneous (SC) injection of AZD2373 dose 1 (6 subjects) or matching placebo (2 subjects).
  Interventions: Drug: AZD2373 subcutaneous injection; Drug: Placebo
- Cohort 2 (Experimental): Once weekly for 6 weeks dosing on Days 1, 8, 15, 22, 29 and 36 randomized subjects will receive a subcutaneous (SC) injection of AZD2373 dose 2 (6 subjects) or matching placebo (2 subjects).
  Interventions: Drug: AZD2373 subcutaneous injection; Drug: Placebo
- Cohort 3 (Experimental): Three times weekly for 6 weeks dosing each week on Days 1, 3, and 5 randomized subjects will receive a subcutaneous (SC) injection of AZD2373 dose 3 (6 subjects) or matching placebo (2 subjects).
  Interventions: Drug: AZD2373 subcutaneous injection; Drug: Placebo
- Cohort 4 (optional) (Experimental): Between one to seven doses each week for 6 weeks randomized subjects will receive a subcutaneous (SC) injection of AZD2373 dose 4 (6 subjects) or matching placebo (2 subjects).
  Interventions: Drug: AZD2373 subcutaneous injection; Drug: Placebo
- Cohort 5 (optional) (Experimental): Between one to seven doses each week for 6 weeks randomized subjects will receive a subcutaneous (SC) injection of AZD2373 dose 5 (6 subjects) or matching placebo (2 subjects).
  Interventions: Drug: AZD2373 subcutaneous injection; Drug: Placebo

INTERVENTIONS:
Drug: AZD2373 subcutaneous injection — Randomized subjects will receive multiple ascending dose of AZD2373 by SC injection (dose 1, dose 2, dose 3, dose 4, dose 5).
Drug: Placebo — Randomized subjects will receive a multiple ascending dose of placebo (saline solution) by SC injection.

SUMMARY:
This is a Phase 1 study to assess the the safety, tolerability and pharmacokinetics (PK) of AZD2373, following subcutaneous (SC) administration of multiple ascending doses (MAD) of AZD2373 in healthy male participants of sub-Saharan West African ancestry.

DETAILED DESCRIPTION:
This study will be conducted as a single center, randomized, placebo-controlled, single-blind study to assess the effect of AZD2373 following multiple ascending dose sequential group design administrations to healthy male participants of sub Saharan West African ancestry.

The study will consist of up to 5 cohorts

Up to 40 male participants aged 18 to 55 years (inclusive), at time of informed consent, will be randomized. The MAD study subjects will be selected based on the results of the pre-screening study with regards to APOL1 allele status.

For all cohorts, 8 participants will participate in each cohort.

The expected duration for any participant participating in the study is approximately 14 to 16 weeks, excluding an up to 35-day Screening Period.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male participants of sub-Saharan West African ancestry aged 18 to 55 years (inclusive, at time of informed consent)
3. Have a BMI between 18.5 and 35 kg/m2 (inclusive) and weigh at least 50 kg and no more than 120 kg (inclusive) at screening.
4. Provision of signed, written and dated informed consent and completed mandatory genotyping in the pre-screening study .

Exclusion Criteria:

1. Participants with known ancestry outside of sub-Saharan West Africa.

2. History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.

3. History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.

4. History of any chronic skin disease, auto-immunological diseases and allergic diseases of any etiology.

5. Any clinically important illness, medical/surgical procedure or trauma within 4 weeks prior to administration of IMP on Study Day 1.

6. Participant has clinical signs and symptoms consistent with SARS-CoV-2 or confirmed infection by appropriate laboratory test within the last 4 weeks prior to screening or on admission.

. 7. Participant who had a severe course of COVID-19.

8. Participant has a positive viral RNA test result for SARS-CoV-2 before randomization.

9. Any laboratory values with the following deviations:

1. ALT or AST greater than ULN and clinically significant as determined by the PI.
2. WBC count < 3.0 x 109/L.
3. Hb below LLN.
4. Total bilirubin > ULN.
5. Platelet count below LLN.

   10, Any clinically important abnormalities in clinical chemistry, hematology or urinalysis results, as judged by the PI.

   11. Any positive result on Screening for serum hepatitis B surface antigen, hepatitis C antibody and HIV.

   12. Any abnormal vital signs, after 10 minutes supine rest.

   13. Any clinically significant abnormalities in rhythm, conduction or morphology of the resting ECG and any clinically significant abnormalities in the 12-lead ECG as considered by the Investigator that may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology.

   14. Known or suspected history of drug abuse as judged by the PI.

   15. Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the previous 3 months.

   16. History of alcohol abuse or excessive intake of alcohol as judged by the PI.

   17. Positive screen for drugs of abuse or cotinine (nicotine) at Screening or admission to the Clinical Unit or positive screen for alcohol on admission to the Clinical Unit prior to administration of the IMP on Study Day 1.

   18. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the PI or history of hypersensitivity to drugs with a similar chemical structure or class to AZD2373.

   19. Excessive intake of caffeine-containing drinks or food as judged by the PI.

   20. Use of any prescribed or non-prescribed medication including antacids, analgesics, herbal remedies, mega-dose vitamins or minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long t½..

   21. Plasma donation within one month of the Screening Visit or any blood donation/blood loss > 500 mL during the 3 months prior to the Screening Visit.

   22. Has received another new chemical entity within 3 months prior to administration of the IMP on Study Day.

   23. Participants who have previously received AZD2373. Participants carrying a G2 allele who were enrolled in the AZD2373 SAD study but did not receive AZD2373 are not excluded.

   24. History of severe infection, chronic or recurrent infectious disease or ongoing febrile illness within 30 days prior to Screening.

   25. Evidence of CKD and/or proteinuria.

   26. Blood dyscrasias with increased risk of bleeding including idiopathic thrombocytopenic purpura and thrombotic thrombocytopenic purpura or symptoms of increased risk of bleeding (frequent bleeding gums or nose bleeds).

   27. Involvement of any AstraZeneca or Clinical Unit employee or their close relatives.

   28. Judgment by the PI that the participant should not participate in the study if they have any ongoing or recent (i.e., during the Screening Period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.

   29. Participants who are vegans or have medical dietary restrictions that would make them unable to comply with the diet provided for the in-house Clinical Unit stays.

   30. Participants who cannot communicate reliably with the PI.

   31. Vulnerable participants, eg, kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

   32. History of Trypanosomiasis or Leishmaniasis.

   33. Participants with a planned visit to a tropical or subtropical region within 10 weeks after administration of the IMP or 5 x t½ of AZD2373 (whichever is longer).

   34. Participants with sickle cell disease will be excluded but not individuals with heterozygous sickle cell trait.

   In addition, any of the following is regarded as a criterion for exclusion from the APOL1 genotyping research (APOL1 genotyping to be assessed during the pre-screening study):

   35. Previous bone marrow transplant.

   36. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the APOL1 genotyping sample collection.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events and/or abnormal findings in vital signs, and/or clinical laboratory assessments and/or physical examination and/or electrocardiogram (ECG) evaluation and/or injection site reactions | Up to 21 weeks (From Screening to Final Visit)
  To assess the safety and tolerability of subcutaneous (SC) multiple ascending dose (MAD) administrations of AZD2373.

SECONDARY OUTCOMES:
AUCinf | Up to 16 weeks (From Visit 2 to Final Visit)
  To characterize the PK of AZD2373 following SC MAD administrations of AZD2373
AUCt | Up to 16 weeks (From Visit 2 to Final Visit)
  To characterize the PK of AZD2373 following SC MAD administrations of AZD2373
AUCτ | Up to 16 weeks (From Visit 2 to Final Visit)
  To characterize the PK of AZD2373 following SC MAD administrations of AZD2373
Cmax | Up to 16 weeks (From Visit 2 to Final Visit)
  To characterize the PK of AZD2373 following SC MAD administrations of AZD2373
tmax | Up to 16 weeks (From Visit 2 to Final Visit)
  To characterize the PK of AZD2373 following SC MAD administrations of AZD2373
t1/2 | Up to 16 weeks (From Visit 2 to Final Visit)
  To characterize the PK of AZD2373 following SC MAD administrations of AZD2373
Percent change in plasma APOL1 protein from baseline | Up to 21 weeks (From Screening to Final Visit)
  To assess the effect of SC MAD administrations of AZD2373 on plasma concentrations of APOL1 protein
APOL1 allele status | Days -35 to -1 (Screening period)
  To determine APOL1 G0, G1, G2 allele genotype status in all study participants

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Brooklyn, Maryland, United States